CLINICAL TRIAL: NCT06560580
Title: Comparative Efficacy of 3% Diquafosol Sodium Eye Drops in Dry Eye Patients Across Age Groups: a Propensity Score-Matched Longitudinal Study
Brief Title: Ditefossol Sodium 3% Eye Drops in Patients With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: zhangyi2024
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease
Keywords: diquafosol sodium; age groups; propensity score matching; longitudinal study; dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older group (Other): Patients were divided into two groups based on age: the younger group (<40 years) and the older group (≥40 years). PSM (1:1) was used to ensure no significant differences in baseline characteristics between the two groups
  Interventions: Drug: 3% Diquafosol Sodium Eye Drops
- Younger group (Other): Patients were divided into two groups based on age: the younger group (<40 years) and the older group (≥40 years). PSM (1:1) was used to ensure no significant differences in baseline characteristics between the two groups
  Interventions: Drug: 3% Diquafosol Sodium Eye Drops

INTERVENTIONS:
Drug: 3% Diquafosol Sodium Eye Drops — Each patient was prescribed 3% (5 mL: 150 mg) diquafosol sodium eye drops [Diquas®, provided by Santen Pharmaceutical (China) Co., Ltd.], recommended to instill one drop six times daily for 3 months. Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.

SUMMARY:
This study aimed to evaluate the efficacy of 3% diquafosol sodium eye drops in treating dry eye disease (DED) across different age groups using a propensity score-matched longitudinal design.

DETAILED DESCRIPTION:
1 ）Participants and Study Design

This prospective clinical trial was conducted following ethical principles and received approval from the Ethics Committee of Tianjin Eye Hospital of China (Approval No.: TJYYLCSYSCLL-2021-25). The study adhered to the tenets of the Declaration of Helsinki, and all patients provided written informed consent after receiving a detailed explanation of the study protocols and the potential consequences associated with participation.

Inclusion Criteria: Patients with Dry Eye Disease (DED) were eligible if they met one of the following criteria:

1. They reported symptoms such as dryness, foreign body sensation, burning, fatigue, discomfort, redness, or fluctuating vision, with a Chinese dry eye questionnaire score (DEQS) ≥7. Additionally, they had either a fluorescein tear breakup time (FBUT) ≤5 s, a non-invasive tear breakup time (NIBUT) <10 s, or a Schirmer I test (without anesthesia) ≤5 mm/5 min.
2. They had dry eye-related symptoms with a Chinese DEQS ≥7. Additionally, they had either FBUT >5 s and ≤10 s, NIBUT between 10 and 12 s, or a Schirmer I test (without anesthesia) >5 mm/5 min and ≤10 mm/5 min. Furthermore, patients were required to have positive fluorescein staining (≥5 spots) for diagnosis.

Exclusion Criteria: Excluded were patients with allergies to any component of the drugs or diagnostic agents used; those who had used 3% diquafosol sodium eye drops within 2 weeks before enrollment; any systemic conditions affecting ocular medication; and corneal disorders preventing diagnostic tests, such as keratitis and corneal dystrophy. The exclusion criteria also included concurrent use of ocular or systemic NSAIDs, steroids, or immunosuppressants; recent use of eye drops; recent physical therapy or ocular surgery; recent contact lens wear; punctual plug treatment; independent ocular diseases requiring additional treatment; and pregnant or breastfeeding women or those planning to become pregnant. All female patients of childbearing age tested negative in a urine pregnancy test before enrollment. If both eyes met the inclusion criteria, the eye with the shorter FBUT was selected. If both eyes had the same FBUT, the right eye was selected.

Patients were divided into two groups based on age: the younger group (<40 years) and the older group (≥40 years). Propensity Score Matching (PSM) (1:1) was used to ensure no significant differences in baseline characteristics between the two groups. The study design aimed to evaluate the efficacy of 3% diquafosol eye drops in patients with dry eye across different age groups. Patients were followed up at baseline (V1), 1 month (V2), and 3 months (V3), with examinations including DEQS, visual acuity (VA), lipid layer thickness, tear meniscus height (TMH), meibomian gland dropout area (MGDA), FBUT, Schirmer I test, and intraocular pressure (IOP).

2） Treatment and Examinations

Each patient was prescribed 3% diquafosol sodium eye drops , to be instilled one drop six times daily for 3 months. Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.

The first visit and follow-up examinations included VA, IOP, FBUT, Schirmer I test, TMH, MGDA, DEQS, and lipid layer thickness. The following sequence was used to avoid interference between the tests:

1. **Dry Eye Questionnaire Score (DEQS)**: DEQS was administered first to assess subjective symptoms of dry eye. Patients completed a questionnaire evaluating discomfort and the impact of dry eyes on daily life, with scores calculated using a standardized DEQS scoring system.
2. Visual Acuity (VA): VA was measured using a 5 m standard Snellen chart and recorded in decimal notation. VA was converted to the Logarithm of the Minimum Angle of Resolution (LogMAR) format for statistical analysis.
3. Lipid Layer Thickness: Lipid layer thickness was evaluated using a LipiView interferometer, based on the principle of white-light interference.
4. Tear Meniscus Height (TMH): TMH was measured using an ocular surface analyzer, which captured images of the tear meniscus at the lower eyelid margin to assess tear volume.
5. Meibomian Gland Dropout Area (MGDA): MGDA was examined using an ocular surface analyzer. Infrared imaging visualized the meibomian glands in the eyelids, and the extent of gland dropout was quantified using ImageJ software.
6. Fluorescein Tear Breakup Time (FBUT): FBUT was measured by instilling fluorescein dye into the conjunctival sac and recording the time from the last blink to the first appearance of a dry spot on the corneal surface using a slit-lamp biomicroscope.
7. Schirmer I Test: Schirmer I test was performed without anesthesia. Standardized Schirmer strips were placed at the junction of the middle and lateral thirds of the lower eyelid margins for 5 min. Wetting length on the strip was measured in millimeters.
8. Intraocular Pressure (IOP): IOP was measured using a non-contact tonometer, which delivered a puff of air to the cornea to calculate the IOP. Three measurements were taken for each eye, and the average IOP was recorded.

By following this sequence and using standardized methods, the study ensured a reliable and reproducible assessment of the efficacy of 3% diquafosol eye drops in patients with dry eyes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were based on the Chinese diagnostic criteria for DED16. Patients with DED were eligible if they met one of the following criteria:

1. They reported symptoms such as dryness, foreign body sensation, burning, fatigue, discomfort, redness, or fluctuating vision, with a Chinese dry eye questionnaire score (DEQS) ≥7. Additionally, they had either a fluorescein tear breakup time (FBUT) ≤5 s, a non-invasive tear breakup time (NIBUT) <10 s, or a Schirmer I test (without anesthesia) ≤5 mm/5 min.
2. They had dry eye-related symptoms with a Chinese DEQS ≥7. Additionally, they had either FBUT >5 s and ≤10 s, NIBUT between 10 and 12 s, or a Schirmer I test (without anesthesia) >5 mm/5 min and ≤10 mm/5 min. Furthermore, patients were required to have positive fluorescein staining (≥5 spots) for diagnosis.

Exclusion Criteria:

Excluded were patients with allergies to any component of the drugs or diagnostic agents used; those who had used 3% diquafosol sodium eye drops within 2 weeks before enrollment; any systemic conditions affecting ocular medication; and corneal disorders preventing diagnostic tests, such as keratitis and corneal dystrophy. The exclusion criteria also included concurrent use of ocular or systemic NSAIDs, steroids, or immunosuppressants; recent use of eye drops; recent physical therapy or ocular surgery; recent contact lens wear; punctal plug treatment; independent ocular diseases requiring additional treatment; and pregnant or breastfeeding women or those planning to become pregnant. All female patients of childbearing age tested negative in a urine pregnancy test prior to enrollment. If both eyes met the inclusion criteria, the eye with the shorter FBUT was selected. If both eyes had the same FBUT, the right eye was selected.

Ages: 23 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Dry Eye Questionnaire Score (DEQS) | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  DEQS was administered first to assess the subjective symptoms of dry eye. Patients were asked to complete a questionnaire that included multiple items evaluating discomfort and the impact of dry eyes on daily life. The scores were calculated using a standardized DEQS scoring system.
Visual Acuity (VA): | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  VA was measured using a 5 m standard Snellen chart and recorded in decimal notation. VA was then converted to the Logarithm of the Minimum Angle of Resolution (LogMAR) format for statistical analysis.
Lipid Layer Thickness: | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  The lipid layer thickness was evaluated using a LipiView interferometer based on the principle of white-light interference.
Tear Meniscus Height (TMH): | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  TMH was measured using an ocular surface analyzer. This device captured images of the tear meniscus at the lower eyelid margin to assess tear volume.
Meibomian Gland Dropout Area (MGDA): | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  MGDA was examined using an ocular surface analyzer (Oculus, Wetzlar, Germany). Infrared imaging was employed to visualize the meibomian glands in the eyelids, and the extent of gland dropout was quantified using the ImageJ software version 1.54j (National Institute of Health, Bethesda, MD, USA).
Fluorescein Tear Breakup Time (FBUT): | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  FBUT was measured by instilling a fluorescein dye into the conjunctival sac and instructing the patient to blink several times to spread the dye uniformly. The time from the last blink to the first appearance of a dry spot on the corneal surface was recorded using a slit-lamp biomicroscope (Nidek. Gamagori, Japan) with a cobalt blue light. The test was performed thrice for each eye, and the average time was calculated.
Schirmer I Test: | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  Schirmer I test was performed without anesthesia. Standardized Schirmer strips were placed at the junction of the middle and lateral thirds of the lower eyelid margins for 5 min. Wetting length on the strip was measured in millimeters to assess basal and reflex tear production. This test was performed at least 30 min after the FBUT test to prevent interference.

SECONDARY OUTCOMES:
Intraocular Pressure (IOP): | Follow-up examinations were conducted at baseline, 1 month, and 3 months after treatment initiation.
  IOP was measured using a non-contact tonometer (Suoer, Zhongshan, China). The device delivered a puff of air to the cornea, and the resistance was used to calculate the IOP. Three measurements were taken for each eye and the average IOP was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Director — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided